CLINICAL TRIAL: NCT01200355
Title: A Randomized Open-Label Trial of Posaconazole Versus Micafungin for Prophylaxis Against Invasive Fungal Infections During Neutropenia in Patients Undergoing Chemotherapy for Acute Myelogenous Leukemia, Acute Lymphocytic Leukemia or Myelodysplastic Syndrome
Brief Title: Posaconazole Versus Micafungin for Prophylaxis Against Invasive Fungal Infections During Neutropenia in Patients Undergoing Chemotherapy for Acute Myelogenous Leukemia, Acute Lymphocytic Leukemia or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-038
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
Keywords: MICAFUNGIN; POSACONAZOLE; antifungal; prolonged neutropenia; 10-038
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Micafungin; posaconazole

ARMS (2):
- micafungin (Experimental): This is a single institution (MSKCC), randomized, open-label comparative trial of micafungin and posaconazole administered as prophylaxis against fungal infections during neutropenia following induction chemotherapy for myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), myelodysplastic syndrome (MDS).
  Interventions: Drug: micafungin
- posaconazole (Experimental): This is a single institution (MSKCC), randomized, open-label comparative trial of micafungin and posaconazole administered as prophylaxis against fungal infections during neutropenia following induction chemotherapy for myelogenous leukemia (AML), acute lymphocytic leukemia (ALL), myelodysplastic syndrome (MDS).
  Interventions: Drug: posaconazole

INTERVENTIONS:
Drug: micafungin — Micafungin 100 mg intravenously once daily. Randomized treatment will be initiated 24-48 h after completion of the last dose of chemotherapy.
  Arms: micafungin
Drug: posaconazole — Posaconazole 400 mg orally twice daily. Randomized treatment will be initiated 24-48 h after completion of the last dose of chemotherapy.
  Arms: posaconazole

SUMMARY:
The purpose of this study is to compare the effects, good and/or bad, of posaconazole and micafungin in preventing fungal infections after chemotherapy for acute leukemia or myelodysplastic syndrome. When people take chemotherapy, they are more likely to get infections. Posaconazole has been approved for the prevention of fungal infections in patients who receive induction chemotherapy for acute leukemia and myelodysplastic syndrome. Posaconazole is available only as an oral suspension and has to be given with food. After chemotherapy, many patients are not able to tolerate food or oral medication because of severe mucositis. Patients unable to tolerate food and oral medications cannot take posaconazole.

Micafungin is an antifungal medication that is given only intravenously. Micafungin is approved for the treatment of certain fungal infections and for preventing fungal infections in patients who receive bone marrow transplant. The investigators know that micafungin is safe. Micafungin has not been tested for the prevention of fungal infections in patients receiving chemotherapy for acute leukemia and myelodysplastic syndrome. Because micafungin is given by vein, it can be given even in patients who cannot take food or medications by mouth after chemotherapy. In this study the investigators want to compare micafungin to posaconazole when given for the prevention of fungal infections in leukemia and myelodysplastic syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of greater than or equal to 18 years of age of either sex and of any race.

Disease definition:

* Anticipated or documented prolonged neutropenia (ANC<500/mm3 [0.5x109/L]) at baseline or likely to develop within 3 to 5 days and lasting for at least 7 days due to:
* Intensive induction chemotherapy for new diagnosis of acute myelogenous leukemia, acute lymphocytic leukemia or myelodysplastic syndrome receiving standard anthracycline based chemotherapy
* Re-induction of acute myelogenous or lymphocytic leukemia after primary relapse
* Myelodysplastic syndromes requiring induction (myelosuppressive) chemotherapy
* Female subjects of childbearing potential must have a negative serum pregnancy test as per MSKCC guidelines.
* Able to swallow oral medications

Exclusion Criteria:

* Subjects with history of presumed or proven invasive fungal infection within 30 days of randomization.
* Subjects who are taking the following:

Drugs known to interact with posaconazole and that may lead to life-threatening side effects (terfenadine, cisapride, and ebastine at entry or within 24 hours before entry, or astemizole at entry or within 10 days before entry); b. Drugs known to lower the serum concentration/efficacy of posaconazole: cimetidine, rifampin, carbamazepine, phenytoin, rifabutin, barbiturates, and isoniazid at entry or within 24 hours before entry; c. Subjects who are planned to receive > 2mg flat dose of vinca alkaloids.

* Subjects with a history of hypersensitivity or idiosyncratic reactions to azole agents.
* Subjects with renal insufficiency (estimated creatinine clearance less than 20 mL/minute at baseline or likely to require dialysis during the study).
* Subjects having an electrocardiogram with a prolonged QTc interval by manual reading: QTc greater than 490 msec.
* Subjects with moderate or severe liver dysfunction at baseline, defined as aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase levels greater than 5 times the upper limit of normal (ULN), or a total bilirubin level greater than 3 times the ULN.
* Subjects who are undergoing re-induction chemotherapy and have participated in this study during their first induction chemotherapy.
* Subjects who will be receiving dasatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2010-09-09 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Genovefa Papanicolaou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Protocol Open to Accrual 09/09/2010 Protocol Closed to Accrual 04/20/2016 Primary Completion Date 04/20/2016 Recruitment Location is the medical clinic
Period: Overall Study
Arm/Group | Micafungin | Posaconazole
Started | 58 | 55
Completed | 51 | 53
Not Completed | 7 | 2
Not completed — Death | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micafungin | Posaconazole | Total
Number analyzed (Participants) | 58 | 55 | 113
Age, Continuous [Median (Full Range); unit: years] | 61 [32 to 75] | 59 [26 to 74] | 61 [32 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 33 | 29 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 5 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 50 | 43 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 58 | 55 | 113

OUTCOME MEASURES:

1. Primary Outcome: Time to Failure
Description: Clinical failure is defined as: 1) need for systemic antifungal therapy (AmBisome) for > 3 consecutive days for presumptive fungal infection, toxicity or intolerance of study medication or 2) death.
Time Frame: 2 years
Population: Analysis based on a modified intention-to-treat (mITT) approach, with the use of data from patients who underwent randomization and received 2 or more doses of prophylaxis. Trial designed w/ power to detect absolute differences of ~25% of prophylaxis failure in the two groups with ~ 80% power and a significance level of 5% using a two-tail test.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Micafungin | Posaconazole
Number analyzed (Participants) | 58 | 55
Days | 16 [12 to 20] | 13 [6 to 16]

2. Secondary Outcome: To Compare the Number of Days on Study Drug Between Patients Who Receive Posaconazole and Patients Who Receive Micafungin.
Time Frame: 2 years
Population: Results reflect patients who discontinued prophylaxis for suspected IFI (invasive fungal infection)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Micafungin | Posaconazole
Number analyzed (Participants) | 58 | 55
days | 11 [8 to 16] | 12 [9 to 14]

3. Secondary Outcome: To Compare the Incidence of Possible, Probable or Proven Invasive Fungal Infections Between Patients Who Receive Posaconazole and Those Who Receive Micafungin During Treatment Phase
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Micafungin | Posaconazole
Number analyzed (Participants) | 58 | 55
Participants | 5 | 3

4. Secondary Outcome: Prophylaxis Failure of Study Medication for Any Reason Between Patients Who Receive Posaconazole and Those Who Receive Micafungin.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Micafungin | Posaconazole
Number analyzed (Participants) | 58 | 55
Participants
  Prophylaxis failure | 20 | 29
  No prophylaxis failure | 38 | 26

5. Secondary Outcome: To Compare Overall Survival Rates at 6 Weeks
Time Frame: 6 weeks from randomization between the two treatment arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Micafungin | Posaconazole
Number analyzed (Participants) | 58 | 55
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Micafungin | Posaconazole
All-Cause Mortality (participants affected / at risk) | 7/58 | 2/55
Serious Adverse Events (participants affected / at risk) | 22/58 | 11/55
Other Adverse Events (participants affected / at risk) | 0/58 | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micafungin (N=58) | Posaconazole (N=55)
Bilirubin Increased (Investigations) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 | 3
Fever (General disorders) | 2 | 2
Gastrointestinal Disorder (Gastrointestinal disorders) | 2 | 0
Immune system disorders - Other, specify (Immune system disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 6 | 2
Multi-organ failure (General disorders) | 1 | 0
Oral Pain (Gastrointestinal disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory infection (Infections and infestations) | 3 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Platelet count decreased (Investigations) | 0 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Blood and lymphatic system disorders - Other, spec (Blood and lymphatic system disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-16): https://cdn.clinicaltrials.gov/large-docs/55/NCT01200355/Prot_SAP_000.pdf